CLINICAL TRIAL: NCT02230592
Title: PET Imaging of Brain mGluR1 Receptors Using [18F]FIMX
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140016; 14-M-0016
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2016-07-18

CONDITIONS: Anxiety Disorder; Major Depressive Disorder
Keywords: PET; Metabolic Glutamate Receptors; Brain Imaging
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Objective:

Metabotropic glutamate receptors (mGluRs) are G-protein coupled receptors that respond to glutamate by activating proteins inside nerve cells that affect cell metabolism, thereby fine-tuning the signals sent between cells to maintain balance in neuronal activity. mGluR subtype 1 (mGluR1s) are located in several brain regions, including the cerebellum, hippocampus, olfactory bulb, and basal ganglia. mGluR1 activation stimulates phospholipase C, resulting in phosphoinositide hydrolysis and increased intracellular calcium levels. Successful development of a positron emission tomography (PET) ligand to image mGlurR1 would impact clinical management of brain disorders characterized by disruptions in glutamatergic transmission, including anxiety and stress disorders, drug addiction, epilepsy, Huntington s disease, and Parkinson s disease. However, detailed study of mGluR1s has heretofore been hindered by the lack of high affinity and selective ligands for this receptor subtype.

The present protocol will evaluate the ability of a new PET ligand, [18F]FIMX, to image and quantify mGluR1 in the brain of healthy human volunteers. This protocol covers four phases:

1. Phase 0: screening whole-body scan;
2. Phase 1: kinetic brain imaging to quantify mGluR1 in brain relative to concurrent measurement of the parent radioligand in arterial plasma;
3. Phase 2: if the tracer is successful in Phase 1, we will estimate radiation-absorbed doses of [18F]FIMX by performing whole body imaging;
4. Phase 3: test-retest analysis of brain binding relative to concurrent measurement of the parent radioligand in arterial plasma.

Study Population:

Healthy adult female and male volunteers (n=22, ages 18 to 55) will undergo brain or whole-body imaging..

Design:

This study will begin with a screening whole-body scan to confirm that the radioactivity has fairly broad distribution in several organs. For absolute quantification of mGluR1, 22 healthy controls will have brain PET imaging using [18F]FIMX and an arterial line. Up to 12 of them will have a test-retest scan. Eight additional subjects will have a whole body PET scan for dosimetry, which does not require an arterial line.

<TAB>

Outcome Measures

To assess absolute quantitation of mGluR1 with [18F]FIMX, we will primarily use two outcome measures: the identifiability and time stability of distribution volume calculated with compartmental modeling. In test-retest study, we will calculate the retest variability. To assess whole-body biodistribution and dosimetry of [18F]FIMX we will use the organ time-activity curves....

DETAILED DESCRIPTION:
Objective:

Metabotropic glutamate receptors (mGluRs) are G-protein coupled receptors that respond to glutamate by activating proteins inside nerve cells that affect cell metabolism, thereby fine-tuning the signals sent between cells to maintain balance in neuronal activity. mGluR subtype 1 (mGluR1s) are located in several brain regions, including the cerebellum, hippocampus, olfactory bulb, and basal ganglia. mGluR1 activation stimulates phospholipase C, resulting in phosphoinositide hydrolysis and increased intracellular calcium levels. Successful development of a positron emission tomography (PET) ligand to image mGlurR1 would impact clinical management of brain disorders characterized by disruptions in glutamatergic transmission, including anxiety and stress disorders, drug addiction, epilepsy, Huntington s disease, and Parkinson s disease. However, detailed study of mGluR1s has heretofore been hindered by the lack of high affinity and selective ligands for this receptor subtype.

The present protocol will evaluate the ability of a new PET ligand, [18F]FIMX, to image and quantify mGluR1 in the brain of healthy human volunteers. This protocol covers four phases:

1. Phase 0: screening whole-body scan;
2. Phase 1: kinetic brain imaging to quantify mGluR1 in brain relative to concurrent measurement of the parent radioligand in arterial plasma;
3. Phase 2: if the tracer is successful in Phase 1, we will estimate radiation-absorbed doses of [18F]FIMX by performing whole body imaging;
4. Phase 3: test-retest analysis of brain binding relative to concurrent measurement of the parent radioligand in arterial plasma.

Study Population:

Healthy adult female and male volunteers (n=22, ages 18 to 55) will undergo brain or whole-body imaging.

Design:

This study will begin with a screening whole-body scan to confirm that the radioactivity has fairly broad distribution in several organs. For absolute quantification of mGluR1, 22 healthy controls will have brain PET imaging using [18F]FIMX and an arterial line. Up to 12 of them will have a test-retest scan. Eight additional subjects will have a whole body PET scan for dosimetry, which does not require an arterial line.

<TAB>

Outcome Measures

To assess absolute quantitation of mGluR1 with [18F]FIMX, we will primarily use two outcome measures: the identifiability and time stability of distribution volume calculated with compartmental modeling. In test-retest study, we will calculate the retest variability. To assess whole-body biodistribution and dosimetry of [18F]FIMX we will use the organ time-activity curves.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 to 55.
* Able to give written informed consent.

EXCLUSION CRITERIA:

* Any current Axis I diagnosis.
* Clinically significant laboratory abnormalities.
* Positive HIV test.
* Unable to have an MRI scan.
* History of neurologic illness or injury with the potential to affect study data interpretation.
* Recent exposure to radiation (i.e. PET from other research) that, when combined with this study, would be above the allowable limits.
* Inability to lie flat on camera bed for at least two hours.
* Pregnancy or breast feeding.
* Able to get pregnant but does not use birth control.
* History of drug or alcohol abuse within 6 months or a history of alcohol or drug dependence (excepting nicotine) within 3 years

Exclusion criteria for the dosimetry subjects are the same as reported above, with the exception of MRI contraindications, because an MRI will not be performed in these subjects.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-11-08; Primary Completion 2016-06-16 (Actual); Study Completion 2016-06-16 (Actual)

PRIMARY OUTCOMES:
Ability to measure mGluR1 in brain | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anwyl R. Metabotropic glutamate receptors: electrophysiological properties and role in plasticity. Brain Res Brain Res Rev. 1999 Jan;29(1):83-120. doi: 10.1016/s0165-0173(98)00050-2. PMID 9974152
- [Background] Battaglia G, Bruno V, Pisani A, Centonze D, Catania MV, Calabresi P, Nicoletti F. Selective blockade of type-1 metabotropic glutamate receptors induces neuroprotection by enhancing gabaergic transmission. Mol Cell Neurosci. 2001 Jun;17(6):1071-83. doi: 10.1006/mcne.2001.0992. PMID 11414795
- [Background] Bordi F, Ugolini A. Group I metabotropic glutamate receptors: implications for brain diseases. Prog Neurobiol. 1999 Sep;59(1):55-79. doi: 10.1016/s0301-0082(98)00095-1. PMID 10416961
- [Derived] Veronese M, Zanotti-Fregonara P, Rizzo G, Bertoldo A, Innis RB, Turkheimer FE. Measuring specific receptor binding of a PET radioligand in human brain without pharmacological blockade: The genomic plot. Neuroimage. 2016 Apr 15;130:1-12. doi: 10.1016/j.neuroimage.2016.01.058. Epub 2016 Feb 2. PMID 26850512
- [Derived] Zanotti-Fregonara P, Xu R, Zoghbi SS, Liow JS, Fujita M, Veronese M, Gladding RL, Rallis-Frutos D, Hong J, Pike VW, Innis RB. The PET Radioligand 18F-FIMX Images and Quantifies Metabotropic Glutamate Receptor 1 in Proportion to the Regional Density of Its Gene Transcript in Human Brain. J Nucl Med. 2016 Feb;57(2):242-7. doi: 10.2967/jnumed.115.162461. Epub 2015 Oct 29. PMID 26514176